CLINICAL TRIAL: NCT03898206
Title: Effects of Breaking up Prolonged Sitting on Postprandial Cardiometabolic Disease Risk Markers in Normal Weight Versus Overweight and Obese South Asian Adults
Brief Title: Effects of Breaking up Prolonged Sitting on Postprandial Cardiometabolic Disease Risk Markers in South Asian Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Bedfordshire (Other)
Responsible Party: Principal Investigator, Daniel Bailey, Senior Lecturer in Health, Nutrition and Exercise, University of Bedfordshire
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2019ISPAR003
Record Dates: First submitted 2019-03-28; First posted 2019-04-01 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Cardiovascular Risk Factor; Cardiovascular Diseases; Diabetes; Physical Activity; Sedentary Lifestyle
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus; Motor Activity; Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prolonged sitting (Experimental): Participants will remain seated for 5 h and instructed to reduce excessive movement, only rising from the chair to void.
  Interventions: Other: Prolonged sitting
- Breaking up sitting with walking breaks (Experimental): Participants will rise from the seated position every 30 min throughout the experimental period to walk on a motorised treadmill at a light intensity walking (as determined during the preliminary test) for 3 min. Participants will start walk on a treadmill at 30 min (so physical activity would be at 30-33 min), 60 min (physical activity will be at 60-63 min), 90 min (physical activity will be at 90-93 min), 120 min (physical activity will be 120-123 min), 150 min (physical activity will be at 150-153 min ), and 180 min (physical activity will be at 180-183 min) in the breakfast postprandial period and 30 min (physical activity will be 30-33 min), 60 min (physical activity will be at 60-63 min), and 90 min (physical activity will be at 90-93 min) in the lunch postprandial period. After performing walking activity, they will return to the seated position.
  Interventions: Other: Breaking up sitting with walking breaks

INTERVENTIONS:
Other: Breaking up sitting with walking breaks — See Breaking up sitting with walking breaks arm description
  Arms: Breaking up sitting with walking breaks
Other: Prolonged sitting — See Prolonged sitting arm description
  Arms: Prolonged sitting

SUMMARY:
The purpose of this study is to examine whether breaking up prolonged sitting with short regular bouts of walking can reduce blood sugar and cholesterol levels after eating, which are risk markers for Type 2 diabetes and heart disease. This study will compare these responses in normal weight versus overweight/obese South Asian adults.

DETAILED DESCRIPTION:
Participants will attend a preliminary testing session where height, weight, body fat and waist circumference will be measured. They will be familiarised with a motorised treadmill that will be used during the experimental visit below and will take part in an exercise test to determine a light-intensity walking speed for the experimental visit.

Participants will then attend two experimental visits in a random order:

1. Prolonged sitting: Participants will remain seated for 5 hours and instructed to reduce excessive movement.
2. Breaking up sitting with walking breaks: Participants will rise from the seated position every 30 minutes throughout the experimental period to walk on a motorised treadmill at a light intensity for 3 minutes. After performing walking activity, they will return to the seated position. In addition, blood sample will be taken at the resting position just before each physical activity bout. The activity breaks will be undertaken on 9 occasions, providing a total of 27 min of light intensity activity.

During each visit, blood pressure will be taken 11 times and blood samples will be taken 10 times. Participants will be given a breakfast and lunch meal to consume.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified South Asian ethnicity.
* Self-report sitting at least 7 hours per day.
* Normal weight, overweight or obese.

Exclusion Criteria:

* Unable to speak and read English.
* Contraindications to performing light-intensity walking.
* Diagnosed cardiovascular disease or diabetes.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2019-02-26 (Actual); Primary Completion 2019-10-25 (Estimated); Study Completion 2020-02-25 (Estimated)

PRIMARY OUTCOMES:
Postprandial glucose | Measured over the 5 hour condition period
  Net incremental area under the curve for each 5 h condition will be calculated for glucose

SECONDARY OUTCOMES:
Postprandial triglycerides | Measured over the 5 hour condition period
  Net incremental area under the curve for each 5 h condition will be calculated for triglycerides
Postprandial insulin | Measured over the 5 hour condition period
  Net incremental area under the curve for each 5 h condition will be calculated for insulin
Blood pressure | Measured over the 5 hour condition period
  Mean systolic and diastolic blood pressure over the 5 h conditions

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bedfordshire, Bedford, Bedfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided